CLINICAL TRIAL: NCT02371135
Title: Metagenomic Evaluation of the Gut Microbiome in Patients With Lynch Syndrome and Other Hereditary Colonic Polyposis Syndromes
Status: Active, not recruiting | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Harvard University (Other); Broad Institute of MIT and Harvard (Other)
Responsible Party: Sponsor
Other Study IDs: 15-016
Record Dates: First submitted 2015-02-19; First posted 2015-02-25 (Estimated); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Lynch Syndrome; Hereditary Colonic Polyposis Syndromes
Keywords: Gut Microbiome; 15-016
MeSH Terms: conditions — Colorectal Neoplasms, Hereditary Nonpolyposis | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — tissue stool

GROUPS / COHORTS (1):
- patients having lower endoscopy: At least 2 weeks prior to scheduled lower endoscopy, consented study participants will be mailed a Brief Diet and Lifestyle Questionnaire, a stool collection kit with detailed instructions and a Stool Collection Data Sheet. No more than one week prior to the lower endoscopy but prior to initiation of bowel preparation, the consented participants will provide a stool specimen and fill out the two questionnaires. The routine lower endoscopy will be performed according to routine clinical procedures. Clinical biopsies of suspicious areas and/or lesions will be taken as per standard clinical care with all such tissue samples sent to pathology for routine clinical analysis. For the sole purposes of research, at the routine lower endoscopy, up to 8 additional colonic biopsies will be taken from normal appearing colon mucosa
  Interventions: Genetic: colonic biopsies; Genetic: questionnaires

INTERVENTIONS:
Genetic: colonic biopsies
Genetic: questionnaires

SUMMARY:
The purpose of this study is to understand the role bacteria that normally live in the colon may play in colorectal cancer risk, in addition to the hereditary risk to colorectal cancer. The investigators will collect stool specimens as well as additional colon biopsy specimens during the patient's scheduled colonoscopy procedure. The investigators will also collect a questionnaire about diet and lifestyle. The samples will be used to study the impact of diet on naturally-occurring oral and gut bacteria and their influences on human health including risk of cancer.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female age 18 or older
* Hereditary colorectal cancer syndrome with one of the following:

  * Lynch syndrome, as defined by the presence of a deleterious germline mutation in the MLH1, MSH2, MSH6, PMS2 or EPCAM genes
  * Other hereditary colonic polyposis syndromes, as defined by the presence of a deleterious germline mutation in any one of the following polyposis genes (APC, biallelic MYH, STK11, SMAD4, BMPR1A, or other CRC-risk associated genes at discretion of PI)

Exclusion Criteria:

* Unable to provide informed consent for testing
* Unable to complete English language questionnaire
* Receiving active chemotherapy
* Having completed active chemotherapy less then 12 months prior to day of scheduled lower endoscopy
* No infectious or drug induced colitis less then 12 months prior to day of scheduled lower endoscopy
* No history of inflammatory colitis (Crohn's disease or ulcerative colitis)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Potential research subjects will be identified prospectively within the clinics of the Clinical Genetics and Gastroenterology Services, of MSKCC.
Sampling Method: Non-Probability Sample
Enrollment: 77 (Actual)
Dates: Start 2015-02 (Actual); Primary Completion 2027-02 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
association of the gut microbiome and dietary factors (To validate said associations, individual questions from the Brief Diet and Lifestyle Questionnaire will be primarily used in the overall analyses) | 2 years
  with risk of adenoma or cancer in Lynch syndrome and other hereditary colonic polyposis syndrome patients. To validate said associations, individual questions from the Brief Diet and Lifestyle Questionnaire will be primarily used in the overall analyses.

CONTACTS AND LOCATIONS:
Overall Officials: Zsofia Stadler, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/